CLINICAL TRIAL: NCT03588806
Title: Use of Xtampza ER to Overcome Difficulties in Swallowing Opioid Pills
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Study halted permanently and will not resume; participants are no longer being examined or receiving intervention.
Sponsor: Ajay Wasan, MD, Msc (Other)
Collaborators: Collegium Pharmaceutical, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Ajay Wasan, MD, Msc, Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: PRO17040444
Record Dates: First submitted 2018-05-07; First posted 2018-07-17 (Actual); Results first posted 2020-06-04 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Chronic Pain; Opioid Use; Deglutition
Keywords: Abuse-deterrent opioid drugs; Xtampza ER
MeSH Terms: conditions — Chronic Pain | interventions — Oxycodone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Xtampza ER (oxycodone) Treatment (Experimental): Following baseline assessments, subjects will have their current opioid medication changed to Xtampza ER (oxycodone) for the duration of the study. A standard conversion table will be used to calculate the dose of Xtampza ER that is equivalent to the subject's current opioid medication dosage. Subjects will be converted to 75% of the calculated dose for the first 7-10 days and then to 100% of the calculated dose for the remaining 3 weeks of the study. The Xtampza ER dosage may be modified at the discretion of the PI to ensure the safety of the subject. As per manufacturer recommendations, subjects will be instructed to open the capsules, sprinkle the microspheres onto soft food such as pudding or applesauce, and then consume the food.
  Interventions: Drug: Xtampza ER (oxycodone)

INTERVENTIONS:
Drug: Xtampza ER (oxycodone) — Following baseline assessments, subjects will have their current opioid medication changed to Xtampza ER (oxycodone) for the duration of the study.

SUMMARY:
This study will examine how the use of Xtampza ER, an opioid analgesic packaged in openable microsphere-containing capsules, affects swallowing satisfaction, pain, and physical and mental health outcomes in chronic pain patients.

DETAILED DESCRIPTION:
An important step in the evolution of pain care is more personalized medicine. One aspect of personalized medicine emphasizes that patients often have additional requirements for prescription medicines beyond just pain relief, including ease in taking medications and overall satisfaction with their care. Surveys indicate that 20% of adult patients either with or without pain have difficulty swallowing their medications, and up to 10% refuse to take a specific therapy because they cannot swallow the pills [1-3]. It is likely that this issue compromises the quantity, quality, and satisfaction with pain relief from oral opioids.

Xtampza ER is an opioid analgesic consisting of a microsphere-containing capsule that can be opened so the microspheres can be added to soft food. This drug is designed to overcome capsule-swallowing issues and therefore may be an important tool for personalized pain medicine care. This study will investigate the pharmaceutic delivery properties of Xtampza to determine whether it is an improved alternative to the pill-swallowing problems that are common with opioid drugs.

ELIGIBILITY:
Inclusion Criteria:

1. Adult subjects must have noncancer chronic pain for at least six months on a daily basis,
2. Be prescribed opioids on a daily basis
3. Have an upper dose limit of daily opioids of 200 mg of morphine equivalents. This is because at doses greater than 200 mg daily, in the investigator's experience it is much more difficult to convert completely to another opioid compound within a week. Fentanyl and methadone users will not be specifically excluded unless their dosages fall outside this range.
4. Ages 21-70
5. Reported difficulty swallowing their opioid medication on the screening form at a level determined significant by the PI.
6. Having a mobile phone. A smart phone is not required to respond to the text messages.
7. Having Internet access to be able to respond to the emailed weekly surveys.
8. If sexually active and able to become pregnant, must agree to use an acceptable method of birth control (hormonal methods, barrier methods with spermicide, intrauterine device (IUD) or abstinence).
9. Only Pain Medicine Clinic patients may participate in this study

Exclusion Criteria:

1. Inability to understand the surveys and complete them.
2. Pregnancy
3. High risk for opioid addiction and/or abuse behaviors
4. Any condition, physical or mental, that in the investigator's judgment precludes optimal participation in the study procedures. This includes any documented current history of liver disease, renal insufficiency, delirium, alcohol use disorder, breast-feeding mothers, acute or severe asthma, chronic obstructive pulmonary disease requiring home oxygen, GI obstruction, biliary tract disease, pancreatitis, cardiac arrhythmia, bladder or urethral obstruction, adrenal insufficiency, psychosis, or taking medications which are potent inhibitors of the CYP3A4 enzyme (such as protease inhibitors, macrolide antibiotics, or antifungals).
5. Demonstration of abusive alcohol behavior. For women, this is more than 3 drinks on any single day or more than 7 drinks per week. For men, more than 4 drinks on any single day or more than 14 drinks per week.
6. Currently taking fentanyl or methadone
7. Exhibiting the following contraindicated conditions: (1) significant respiratory depression (2) acute or severe bronchial asthma in an unmonitored setting or in the absence of resuscitative equipment (3) known or suspected gastrointestinal obstruction, including paralytic ileus (4) hypersensitivity (e.g. anaphylaxis) to oxycodone (5) patients with chronic pulmonary disease (6) elderly, cachet, or debilitated patients (7) patients with evidence of increased intracranial pressure, brain tumors, head injury, or impaired consciousness (8) patients with seizure disorders (9) pregnant and breastfeeding women, due to risks to the fetus/baby

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2019-07-31 (Actual); Study Completion 2019-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ajay D Wasan, MD, MSc, Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Pain Medicine at Centre Commons, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fields J, Go JT, Schulze KS. Pill Properties that Cause Dysphagia and Treatment Failure. Curr Ther Res Clin Exp. 2015 Aug 20;77:79-82. doi: 10.1016/j.curtheres.2015.08.002. eCollection 2015 Dec. PMID 26543509
- [Background] Engelhard E, Smith C, Vervoort S, Kroon F, Brinkman K, Nieuwkerk P, Reiss P, Geerlings S. Patients' willingness to take separate component antiretroviral therapy regimens for HIV in the Netherlands. J Int AIDS Soc. 2014 Nov 2;17(4 Suppl 3):19536. doi: 10.7448/IAS.17.4.19536. eCollection 2014. PMID 25394045
- [Background] Llorca PM. Discussion of prevalence and management of discomfort when swallowing pills: orodispersible tablets expand treatment options in patients with depression. Ther Deliv. 2011 May;2(5):611-22. doi: 10.4155/tde.11.32. PMID 22833978
- [Background] Pergolizzi JV Jr, Taylor R Jr, Nalamachu S, Raffa RB, Carlson DR, Varanasi RK, Kopecky EA. Challenges of treating patients with chronic pain with dysphagia (CPD): physician and patient perspectives. Curr Med Res Opin. 2014 Feb;30(2):191-202. doi: 10.1185/03007995.2013.854197. Epub 2013 Oct 28. PMID 24117419
- [Background] Deyo RA, Dworkin SF, Amtmann D, Andersson G, Borenstein D, Carragee E, Carrino J, Chou R, Cook K, DeLitto A, Goertz C, Khalsa P, Loeser J, Mackey S, Panagis J, Rainville J, Tosteson T, Turk D, Von Korff M, Weiner DK. Report of the NIH Task Force on research standards for chronic low back pain. J Pain. 2014 Jun;15(6):569-85. doi: 10.1016/j.jpain.2014.03.005. Epub 2014 Apr 29. PMID 24787228
- [Background] Wasan AD, Michna E, Edwards RR, Katz JN, Nedeljkovic SS, Dolman AJ, Janfaza D, Isaac Z, Jamison RN. Psychiatric Comorbidity Is Associated Prospectively with Diminished Opioid Analgesia and Increased Opioid Misuse in Patients with Chronic Low Back Pain. Anesthesiology. 2015 Oct;123(4):861-72. doi: 10.1097/ALN.0000000000000768. PMID 26375824
- [Background] Jamison RN, Ross EL, Michna E, Chen LQ, Holcomb C, Wasan AD. Substance misuse treatment for high-risk chronic pain patients on opioid therapy: a randomized trial. Pain. 2010 Sep;150(3):390-400. doi: 10.1016/j.pain.2010.02.033. Epub 2010 Mar 23. PMID 20334973
- [Background] Wasan AD, Davar G, Jamison R. The association between negative affect and opioid analgesia in patients with discogenic low back pain. Pain. 2005 Oct;117(3):450-461. doi: 10.1016/j.pain.2005.08.006. PMID 16154274

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Xtampza ER (Oxycodone) Treatment
Started | 11
Completed | 11
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Xtampza ER (Oxycodone) Treatment
Number analyzed (Participants) | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 11
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.5 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 11
Daily Pain Intensity [Mean (Standard Deviation); unit: units on a scale] — Daily Pain Intensity is a measure of how intense an individual's pain was in the last 24 hours on a 0-10 scale, with 0 meaning "no pain" and 10 meaning "the worst pain imaginable." Higher scores indicate higher pain levels.
  units on a scale | 8.1 (1.7)
Weekly Pain Intensity [Mean (Standard Deviation); unit: units on a scale] — Weekly Pain Intensity is a measure of how intense an individual's pain was in the last 7 days on a 0-10 scale, with 0 meaning "no pain" and 10 meaning "the worst pain imaginable." Higher scores indicate higher pain levels.
  units on a scale | 8.0 (2.0)
Swallowing Difficulty [Mean (Standard Deviation); unit: units on a scale] — Pill swallowing difficulty is a measure of how much difficulty an individual has swallowing pills on a 0-10 scale with 0 being "no trouble at all" and 10 being "the greatest difficulty possible." Higher scores indicate greater swallowing difficulty.
  units on a scale | 6.7 (1.8)
Opioid medication satisfaction [Mean (Standard Deviation); unit: units on a scale] — Opioid medication satisfaction is a measure of how satisfied an individual is with their current opioid medication on a 0-10 scale with 0 being "not satisfied at all" and 10 being "completely satisfied." Higher scores indicate higher satisfaction.
  units on a scale | 4.3 (2.8)

OUTCOME MEASURES:

1. Primary Outcome: Effect of Xtampza ER Conversion on Pain Intensity in the Last 24 Hours
Description: Percent change in pain intensity (in the last 24 hours) from baseline to the end of the study averaged over the last 7 days before clinic visit 4 (week 6). Pain Intensity is measured on a 0-10 scale, with 0 meaning "no pain" and 10 meaning "the worst pain imaginable." As decreases in pain intensity are a sign of improvement, percent change in pain intensity is calculated as -(end of study - baseline)/baseline score.
Time Frame: Measured at baseline and at the end of the 6-week study
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Xtampza ER (Oxycodone) Treatment
Number analyzed (Participants) | 11
percent change | 12.5 (31.5)
Statistical Analysis 1: Comparison: Xtampza ER (Oxycodone) Treatment; Test type: Superiority; p = 0.218, ANOVA; Univariate repeated measures ANOVA

2. Primary Outcome: Effect of Xtampza ER Conversion on Pain Intensity in the Last 7 Days
Description: Percent change in pain intensity (in the past 7 days) from baseline to the end of the study at clinic visit 4 (week 6). Pain Intensity is measured on a 0-10 scale, with 0 meaning "no pain" and 10 meaning "the worst pain imaginable." As decreases in pain intensity are a sign of improvement, percent change in pain intensity is calculated as -(end of study - baseline)/baseline score.
Time Frame: Measured at baseline and at the end of the 6-week study
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Xtampza ER (Oxycodone) Treatment
Number analyzed (Participants) | 11
percent change | 9.3 (30)
Statistical Analysis 1: Comparison: Xtampza ER (Oxycodone) Treatment; Test type: Superiority; p = 0.268, ANOVA; Univariate repeated measures

3. Secondary Outcome: Change in Pill Swallowing Difficulty Score
Description: Pill swallowing difficulty will be measured via a 0-10 scale with 0 being "no trouble at all" and 10 being "the greatest difficulty possible." Responses will be summarized as change from baseline scores to the end of the study at clinic visit 4 (week 6).
Time Frame: Measured at baseline and at the end of the 6-week study. Baseline covers current opioid medication, and week 6 covers Xtampza ER.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Xtampza ER (Oxycodone) Treatment
Number analyzed (Participants) | 11
units on a scale | -5.7 (2.6)
Statistical Analysis 1: Comparison: Xtampza ER (Oxycodone) Treatment; Test type: Superiority; p < 0.001, ANOVA; Univariate repeated measures ANOVA

4. Secondary Outcome: Patient-Reported Outcomes Measurement Information System (PROMIS) Pain Interference
Description: The Pain Interference questions (#25-28) from the PROMIS-29 Adult Profile v2.0. Questions are measured on a 5-point scale with 1 being "Not at all" and 5 being "Very much". Responses will be summed and converted to T-Scores using the Assessment Center PROMIS Scoring Service (www.assessmentcenter.net), which rescales the raw score to a standardized T-Score with a population mean of 50 and standard deviation of 10. Pain Interference T-Scores will be summarized as the change from baseline scores to the end of the study at clinic visit 4 (week 6).
Time Frame: Measured at baseline and at the end of the 6-week study
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | Xtampza ER (Oxycodone) Treatment
Number analyzed (Participants) | 11
T-Score | -3.6 (8.2)
Statistical Analysis 1: Comparison: Xtampza ER (Oxycodone) Treatment; Test type: Superiority; p = 0.228, ANOVA; Univariate repeated measures ANOVA

5. Secondary Outcome: Opioid Medication Satisfaction
Description: Opioid medication satisfaction will be measured via a 0-10 scale with 0 being "not satisfied at all" and 10 being "completely satisfied." Responses will be summarized as change from baseline score to the end of the study at clinic visit 4 (week 6).
Time Frame: Measured at baseline and at the end of the 6-week study. Recorded baseline for current opioid medication and in week 6 for Xtampza ER.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Xtampza ER (Oxycodone) Treatment
Number analyzed (Participants) | 11
units on a scale | 2.8 (4.0)
Statistical Analysis 1: Comparison: Xtampza ER (Oxycodone) Treatment; Test type: Superiority; p = 0.043, ANOVA; Univariate repeated measures ANOVA

6. Secondary Outcome: PROMIS Depression, Anxiety, Satisfaction With Social Roles, and Sleep Disturbance
Description: The Depression (#9-12), Anxiety (#5-8), Satisfaction with Social Roles (#21-24), and Sleep Disturbance (#17-20) questions from the PROMIS-29 Adult Profile v2.0. Questions are measured on a 5-point scale with 1 being "Never" and 5 being "Always". Responses for each section will be summed and converted to T-Scores using the Assessment Center PROMIS Scoring Service (www.assessmentcenter.net), which rescales the raw score to a standardized T-Score with a population mean of 50 and standard deviation of 10. These T-Scores will be summarized as change from baseline scores to the end of the study at clinic visit 4 (week 6).
Time Frame: Measured at baseline and at the end of the 6-week study
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | Xtampza ER (Oxycodone) Treatment
Number analyzed (Participants) | 11
T-Score
  Depression | -0.4 (7.3)
  Anxiety | -1.7 (6.1)
  Satisfaction with Social Roles | 1.1 (4.9)
  Sleep Disturbance | -3.7 (6.2)
Statistical Analysis 1: Comparison: Xtampza ER (Oxycodone) Treatment; PROMIS Social Roles score; Test type: Superiority; p = 0.486, ANOVA; Univariate repeated measures ANOVA
Statistical Analysis 2: Comparison: Xtampza ER (Oxycodone) Treatment; PROMIS Sleep Disturbance T-Scores; Test type: Superiority; p = 0.078, ANOVA; Univariate repeated measures ANOVA
Statistical Analysis 3: Comparison: Xtampza ER (Oxycodone) Treatment; PROMIS Depression T-Scores; Test type: Superiority; p = 0.874, ANOVA; Univariate repeated measures ANOVA
Statistical Analysis 4: Comparison: Xtampza ER (Oxycodone) Treatment; PROMIS Anxiety T-Score; Test type: Superiority; p = 0.389, ANOVA; Univariate repeated measures ANOVA

7. Secondary Outcome: PROMIS Physical Function
Description: The Physical Function questions (#1-4) from the PROMIS-29 Adult Profile v2.0. Questions are measured on a 5-point scale with 5 being "Without any difficulty" and 1 being "Unable to do". Responses will be summed and converted to T-Scores using the Assessment Center PROMIS Scoring Service (www.assessmentcenter.net), which rescales the raw score to a standardized T-Score with a population mean of 50 and standard deviation of 10. Physical Function T-Scores will be summarized as change from baseline score to the end of the study at clinic visit 4 (week 6).
Time Frame: Measured at baseline and at the end of the 6-week study
Measure: Mean (Standard Deviation); unit: T-Score
Arm/Group | Xtampza ER (Oxycodone) Treatment
Number analyzed (Participants) | 11
T-Score | 0.7 (5.0)
Statistical Analysis 1: Comparison: Xtampza ER (Oxycodone) Treatment; Test type: Superiority; p = 0.676, ANOVA; Univariate repeated measures ANOVA

8. Secondary Outcome: Patient Global Impression of Change (PGIC)
Description: The subject's impression of the impact of the treatment on their pain and function will be measured with a 7-item scale (-3 = very much worse, -2 = much worse, -1 = minimally worse, 0 = no change, 1 = minimally improved, 2 = much improved, 3 = very much improved). Responses will be summarized as individual mean scores at clinic visit 4 (week 6).
Time Frame: Recorded in week 6.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Xtampza ER (Oxycodone) Treatment
Number analyzed (Participants) | 11
units on a scale | 1.2 (1.1)

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: Standard definitions of adverse and/or serious adverse events were used.
Arm/Group | Xtampza ER (Oxycodone) Treatment
All-Cause Mortality (participants affected / at risk) | 0/11
Serious Adverse Events (participants affected / at risk) | 0/11
Other Adverse Events (participants affected / at risk) | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2018-02-09): https://cdn.clinicaltrials.gov/large-docs/06/NCT03588806/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2017-11-10): https://cdn.clinicaltrials.gov/large-docs/06/NCT03588806/Prot_SAP_001.pdf